CLINICAL TRIAL: NCT06706713
Title: An Apen-label, Multicenter Phase II Study to Evaluate the Efficacy and Safety of BEBT-109 in Patients With EGFR Exon 20 Insertion Mutations in Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Study of BEBT-109 in Subjects With EGFR Exon 20 Insertion Mutations Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BeBetter Med Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBMT-109-P02
Record Dates: First submitted 2024-11-25; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Non-Small Cell Lung Cancer; EGFR Exon 20 Insertion Mutation
Keywords: BEBT-109; EGFR Exon 20 Insertion Mutations; Efficacy; Safety
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: This study is designed with two cohorts, each comprising approximately 100 subjects. Subjects receive BEBT-109 capsules treatment with a dosage of 120mg bid (twice a day), and each 28-day period constitutes a cycle. In case of intolerance during the treatment, dose adjustments can be made according to the adjustment plan.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BEBT-109 Capsule Treatment (Experimental): BEBT-109 Capsule: Administration and dosage: Oral administration, 120mg; Frequency and duration of administration: Twice a day,and 28 days as a treatment cycle.
  Interventions: Drug: BEBT-109 Capsule

INTERVENTIONS:
Drug: BEBT-109 Capsule — Take orally before breakfast and dinner each day, with a minimum interval of 9 hours between doses, 120mg each time, twice a day,and 28 days as a treatment cycle.
  Other Names: KCBT-1083

SUMMARY:
This study is an open-label, multicenter Phase II trial, planning to enroll 200 subjects, using BEBT-109 capsules as monotherapy, aimed at evaluating the efficacy and safety of BEBT-109 capsules in subjects with Epidermal Growth Factor Receptor (EGFR) exon 20 insertion mutations in locally advanced or metastatic Non-Small Cell Lung Cancer （NSCLC）.

DETAILED DESCRIPTION:
This study is designed with two cohorts, each comprising approximately 100 subjects. Cohort 1 includes subjects with EGFR exon 20 insertion mutations in NSCLC who have failed or are intolerant to at least one systemic chemotherapy and have not received third-generation EGFR (Tyrosine Kinase Inhibitor) TKI therapy. Cohort 2 includes subjects with EGFR exon 20 insertion mutations in NSCLC who have failed or are intolerant to at least one systemic chemotherapy and have experienced Progressive Disease after receiving standard-dose third-generation EGFR TKI therapy.Subjects receive BEBT-109 capsules treatment with a dosage of 120mg bid (twice a day), and each 28-day period constitutes a cycle. In case of intolerance during the treatment, dose adjustments can be made according to the adjustment plan.

Each subject's study process includes three phases: the screening period, the treatment period, and the post-treatment follow-up period. The screening period can last up to 28 days.During the treatment period, tumor assessments are conducted every 8 weeks (±7 days). If the initial response is Partial Response (PR) or Complete Response (CR ), a confirmation assessment for efficacy is required between 4-6 weeks. Subjects can continue to receive study medication until Progressive Disease (PD), death, intolerable toxicity occurs, or the subject withdraws informed consent (whichever comes first). After discontinuing treatment, subjects will enter the post-treatment follow-up period, receiving efficacy follow-ups every 8 weeks (±7 days) (until tumor progression or other anti-tumor treatments are administered) and survival follow-ups every 3 months (±7 days).

When a subject experiences the first instance of Progressive Disease, if the investigator believes that continued use of the study medication may still be beneficial, the subject is allowed to continue receiving study medication until imaging indicates no clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have been fully informed and are willing to sign the informed consent form.
2. Age of at least 18 years, with no gender restrictions.
3. According to the 8th edition of the American Joint Committee on Cancer (AJCC) lung cancer Tumor Node Metastasis (TNM) staging criteria: histologically or cytologically confirmed locally advanced (stages IIIB or IIIC, and deemed unsuitable for surgery or radiotherapy by the investigator) or metastatic (stage IV) NSCLC.
4. Written test reports confirm the occurrence of EGFR exon 20 insertion mutations.
5. Cohort 1 includes NSCLC patients who have failed or are intolerant to at least one systemic chemotherapy (defined as having undergone at least one platinum-based chemotherapy regimen or other chemotherapy regimen) and have not received third-generation EGFR TKI treatment; Cohort 2 includes NSCLC patients who have failed or are intolerant to at least one systemic chemotherapy (defined as having undergone at least one platinum-based chemotherapy regimen or other chemotherapy regimen) and have experienced Progressive Disease after receiving standard doses of third-generation EGFR TKI (such as osimertinib 80 mg once daily, or savolitinib 80 mg once daily, or alectinib 110 mg once daily, etc.).
6. Eastern Cooperative Oncology Group (ECOG) score of 0-2, with no decline in physical performance in the past two weeks, and an expected survival of at least 12 weeks.
7. Subjects must have at least one measurable lesion according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 criteria.
8. Laboratory tests indicate that subjects have adequate organ function: including: a. Absolute neutrophil count (ANC) ≥1.5×10^9/L; platelet count (PLT) ≥100×10^9/L; hemoglobin (HGB) ≥80g/L; b. Serum total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN), aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤2.5 times ULN (for those with liver metastasis, total bilirubin ≤3 times ULN, AST and ALT ≤5 times ULN are allowed); c. Creatinine ≤1.5 times ULN, when creatinine >1.5 times ULN, creatinine clearance must be confirmed, and creatinine clearance must be ≥45 ml/min (actual value, or calculated by the Cockcroft-Gault formula); d. Activated partial thromboplastin time (APTT) ≤1.5 times ULN, prothrombin time (PT) ≤1.5 times ULN, international normalized ratio (INR) ≤1.5 times ULN.
9. If the subject is a female with childbearing potential, she must use adequate contraceptive measures (such as condoms), must not breastfeed, and must have a negative blood pregnancy test before dosing.
10. male subjects must be willing to use barrier contraceptive measures during the study period, i.e., condoms.

Exclusion Criteria:

1. Individuals who have had other malignant tumors within 5 years prior to enrollment, except for basal cell carcinoma of the skin that has been removed and cured, in situ bladder cancer, or in situ cervical cancer.
2. Those who have previously received drugs for EGFR exon 20 insertion mutations, such as Poziotinib, Tarloxotinib, TAK788, JNJ-61186372, CLN-081, or high-dose third-generation EGFR TKIs (Osimertinib > 80 mg/day, Furmonertinib > 80 mg/day, or Almonertinib > 110 mg/day, etc.).
3. Any other anti-cancer treatment within 4 weeks prior to the first use of the study drug (including cytotoxic chemotherapy, radiotherapy, immunotherapy, or other biological therapies; for Mitomycin or Nitrosoureas, within 6 weeks; for small molecule targeted drugs, at least 2 weeks or at least 5 half-lives from the last dose, whichever is longer).
4. Received medication from another clinical trial within 4 weeks prior to the first administration of the study treatment.
5. Undergone major surgery (excluding vascular access procedures) within 4 weeks prior to the first administration of the study treatment.
6. Currently using or having used within 1 week known strong inhibitors or inducers of CYP3A4 and CYP2C8, including medications or herbal supplements.
7. At the start of the study treatment, unresolved toxicities from previous treatments that are more than Grade 1 according to the Common Terminology Criteria for Adverse Events (CTCAE), except for alopecia, and neurotoxicity related to previous platinum treatment can be relaxed to Grade 2.
8. Spinal cord compression, meningeal metastasis, or brain metastasis, except for those who are asymptomatic, stable, and have not required steroid medication within 4 weeks prior to the start of the study treatment.
9. Patients with symptomatic and unstable pleural effusion or ascites.
10. Those with severe or uncontrolled systemic diseases requiring treatment, deemed unsuitable for the trial by the investigator, including hypertension, diabetes, chronic heart failure (New York Heart Association (NYHA) class III-IV), unstable angina, myocardial infarction within 1 year, active bleeding, etc..
11. Individuals with uncontrolled active infections.
12. Clinically significant active infections, including Hepatitis B (HBV) and Hepatitis C (HCV). Active Hepatitis B is defined as Hepatitis B surface antigen (HBsAg) positive with detectable HBV DNA copies above the upper limit of normal of the testing laboratory. Patients with HBV DNA copies above the normal limit are allowed to receive antiviral treatment before screening to reduce the viral load to below the normal limit, but must continue antiviral treatment for Hepatitis B during the trial; Active Hepatitis C is defined as HCV RNA above the detection limit.
13. History of immunodeficiency, including positive Human Immunodeficiency Virus (HIV) antibody tests, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
14. At rest, the average corrected QT interval (QTc) from three Electrocardiogram (ECG) examinations is >450 msec (only if the first ECG suggests QTc >450 msec, two more measurements are required, and the average of the three values is taken).
15. Various severe and clinically significant cardiac rhythm, conduction, and resting ECG morphological abnormalities, such as complete left bundle branch block, third-degree block, second-degree block, PR interval >250 msec, etc..
16. Various factors that may increase the risk of QTc prolongation or arrhythmic events, such as heart failure, hypokalemia (low potassium levels indicated in the screening period blood chemistry, except for those who have been treated with potassium supplements and rechecked as normal before the first dose), congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death before the age of 40.
17. History of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active interstitial lung disease.
18. Uncontrollable nausea and vomiting, chronic gastrointestinal disease, inability to swallow drug formulations, or previous extensive bowel resection, which may affect the adequate absorption of BEBT-109.
19. History of hypersensitivity reaction to excipients in the BEBT-109 formulation.
20. Female subjects who are breastfeeding.
21. The investigator determines that the subject has any clinical or laboratory examination abnormalities or other reasons that make them unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR | Every 8 weeks,assessed up to 24 months.
  Objective Response Rate
PFS | Every 8 weeks,assessed up to 24 months.
  Progression-Free Survival

SECONDARY OUTCOMES:
DOR | Every 8 weeks,assessed up to 24 months.
  Duration of Response
DCR | Every 8 weeks,assessed up to 24 months.
  Disease Control Rate
TTR | Every 8 weeks,assessed up to 24 months.
  Time to Response
OS | From date of administration until date of death from any cause, assessed up to 24 months.
  Overall Survival
Adverse Events | From the first dose of medication to 30 days after the last dose in subjects.
  Safety and tolerability are assessed through imaging examinations, systemic adverse events, and laboratory abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Nong Yang, Phd, Principal Investigator — Hunan Cancer Hospital; Yilong Wu, Phd, Principal Investigator — Guangdong Provincial People's Hospital
Locations (2):
- China (2):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan